CLINICAL TRIAL: NCT02009527
Title: Effect of Arginase Inhibition on Endothelial Function Induced by Ischemia-reperfusion in Patients With Coronary Artery Disease
Brief Title: Arginase Inhibition in Ischemia-reperfusion Injury
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, John Pernow, Professor, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: AIR
Record Dates: First submitted 2013-12-08; First posted 2013-12-12 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Coronary Artery Disease; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus, Type 2 | interventions — N(omega)-hydroxynorarginine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- N-hydroxy-nor-arginine (Experimental): N-hydroxy-nor-arginine 0.1 mg/ min i.a. for 20 min
  Interventions: Drug: N-hydroxy-nor-arginine
- NaCl (Placebo Comparator): NaCl 0.9%, 6 ml/min i.a. for 20 min
  Interventions: Drug: NaCl

INTERVENTIONS:
Drug: N-hydroxy-nor-arginine
  Arms: N-hydroxy-nor-arginine
Drug: NaCl
  Arms: NaCl

SUMMARY:
The present project is designed to test the hypothesis that arginase contributes to endothelial dysfunction induced by ischemia-reperfusion in patients with coronary artery disease.

DETAILED DESCRIPTION:
Background: Arginase competes with nitric oxide synthase for their common substrate L-arginine. Up-regulation of arginase in coronary artery disease (CAD) and diabetes mellitus may reduce nitric oxide bioavailability contributing to endothelial dysfunction and ischemia-reperfusion injury. Arginase inhibition reduces infarct size in animal models. Therefore the aim of the current study was to investigate if arginase inhibition protects from endothelial dysfunction induced by ischemia-reperfusion in patients with CAD with or without type 2 diabetes.

Methods: Male patients with CAD (n=12) or CAD + type 2 diabetes (n=12), were included in this cross-over study with blinded evaluation. Endothelium-dependent vasodilatation was assessed by flow-mediated dilatation (FMD) of the radial artery before and after 20 min ischemia-reperfusion during intra-arterial infusion of the arginase inhibitor (N-hydroxy-nor-L-arginine, 0.1 mg/min) or saline.

Results: The forearm ischemia-reperfusion was well tolerated. Endothelium-independent vasodilatation was assessed by sublingual nitroglycerin. Ischemia-reperfusion decreased FMD in patients with CAD from 12.7±5.2% to 7.9±4.0% during saline administration (P<0.05). N-hydroxy-nor-L-arginine administration prevented the decrease in FMD in the CAD group (10.3±4.3% at baseline vs. 11.5±3.6% at reperfusion). Ischemia-reperfusion did not significantly reduce FMD in patients with CAD + type 2 diabetes. However, FMD at reperfusion was higher following nor-NOHA than following saline administration in both groups (P<0.01). Endothelium-independent vasodilatation did not differ between the occasions.

Conclusions: Inhibition of arginase protects against endothelial dysfunction caused by ischemia-reperfusion in patients with CAD. Arginase inhibition may thereby be a promising therapeutic strategy in the treatment of ischemia-reperfusion injury.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease

Exclusion Criteria:

* Age >80 years, Myocardial infarction/unstable angina within 6 weeks prior to the study, Raynaud's phenomenon, peripheral vasculopathies, arterial shunting or other vascular surgery of the study arm, Any concomitant disease or condition that may interfere with the possibility for the patient to comply with or complete the study protocol, Participant in an ongoing study, Unwillingness to participate following oral and written information.

Max Age: 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-01; Primary Completion 2013-04 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in endothelial function | 20 min of reperfusion
  Flow-mediated dilatation of the radial artery

CONTACTS AND LOCATIONS:
Overall Officials: John Pernow, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

REFERENCES:
- [Derived] Kovamees O, Shemyakin A, Pernow J. Effect of arginase inhibition on ischemia-reperfusion injury in patients with coronary artery disease with and without diabetes mellitus. PLoS One. 2014 Jul 29;9(7):e103260. doi: 10.1371/journal.pone.0103260. eCollection 2014. PMID 25072937